CLINICAL TRIAL: NCT02707393
Title: Allogeneic Stem Cell Transplantation for Children and Adolescents With CML: Conditioning Regimen, Donor Selection, Supportive Care and Diagnostic Procedures
Brief Title: Allogeneic Stem Cell Transplantation for Children With CML
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Anna Kinderkrebsforschung (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2008-000569-50
Record Dates: First submitted 2016-03-01; First posted 2016-03-14 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: stem cell transplantation; pediatrics
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — fludarabine; fludarabine phosphate; Thiotepa; Melphalan; thymoglobulin; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): Fludarabine intravenous - daily dose: 40mg/sqm on day -7, -6, -5, -4; Thiotepa intravenous - daily dose: 2 x 5mg/kg on day -3; Melphalan intravenous - daily dose: 140/mg/sqm on day - 2; ATG intravenous - dose according to local standards on day -3, -2, -1; bone marrow or peripheral blood stem cells of an HLA identical sibling or matched unrelated donor on day 0; GvHD propyhlaxis with Mycophenolate Mofetil and Cyclosporine A
  Interventions: Drug: Fludarabine; Drug: Thiotepa; Drug: Melphalan; Drug: ATG; Drug: Cyclosporine A; Drug: Mycophenolate mofetil; Biological: bone marrow or peripheral blood stem cells

INTERVENTIONS:
Drug: Fludarabine — infusion
  Other Names: Fludara
Drug: Thiotepa — infusion
  Other Names: Thioplex; TESPA
Drug: Melphalan — infusion
  Other Names: Alkeran
Drug: ATG — infusion
  Other Names: Thymoglobulin
Drug: Cyclosporine A — infusion, orally if possible
  Other Names: Sandimmune
Drug: Mycophenolate mofetil — infusion
  Other Names: CellCept
Biological: bone marrow or peripheral blood stem cells — infusion

SUMMARY:
In children and adolescents with chronic myeloid leukaemia (CML) stem cell transplantation (SCT) may be a valid alternative to the life-long treatment with tyrosinkinase inhibitors (TKI). This trial aims to evaluate the use of a reduced intensity conditioning regimen (RIC), consisting of fludarabine, melphalan and thiotepa in order to minimize transplant related mortality and toxic late effects. Strict post-transplant monitoring and reintroduction of TKI as well as donor lymphocyte infusions (DLI) in case of relevant residual disease are part of the protocol.

DETAILED DESCRIPTION:
Chronic myeloid leukaemia (CML) is a rare disease in children with an incidence of 3-5% of all paediatric leukaemias. Since the introduction of tyrosinkinase inhibitors (TKI) stem cell transplantation (SCT) is no longer the first choice treatment for patients with early phase CML.

However life-long treatment with TKI may not be feasable in several cases due to side effects such as growth retardation, non-compliance and resistance. This protocol evaluates the feasibility of SCT following a reduced intensity conditioning regimen (RIC) consisting of fludarabine, melphalan, thiotepa and thymoglobuline (ATG). Matched siblings and matched unrelated donors are permitted for stem cell donation. In case of unrelated donors tissue typing has to be done by high resolution molecular typing. Donors with 10/10 or 9/10 identical allels in the human leukocyte antigen (HLA) system are accepted. Preferred stem cell source is bone marrow but peripheral blood stem cells and umbilical cord blood are also allowed. Graft-versus-Host-Disease (GvHD)-prophylaxis is achieved with cyclosporine A and mycophenolate mofetil.

Monitoring of the breakpoint cluster region - Abelson (BCR/ABL) rearrangement is performed monthly in the first year after SCT. In case of BCR/ABL positivity TKI are given in the first year after SCT. Followed by donor lymphocyte infusions (DLI) later on if BCR/ABL positivity persists.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents with BCR/ABL positive CML in chronic phase, who are eligible for allogeneic stem cell transplantation, irrespective of the previous treatment strategy
* availability of a HLA matched sibling donor (MSD), a matched family donor, a matched unrelated donor or a matched unrelated cord blood (MD)
* informed consent

Exclusion Criteria:

* unavailability of MSD or MD
* patients in accelerated phase or blast crisis
* pregnancy
* previous autologous or allogeneic SCT
* no informed consent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
transplant related mortality | one year

SECONDARY OUTCOMES:
overall survival | five years
event free survival | five years

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Matthes, MD, Study Chair — St. Anna Kinderspital
Locations (4):
- Austria (2):
  - Universitätsklinik für Kinder- und Jugendheilkunde, Graz
  - St. Anna Kinderspital, Vienna
- Hospital Motol, Department of Pediatric Hematology and Oncology, BMT Unit, Prague, Czechia
- Clinica Pediatrica, Monza, Italy

IPD SHARING:
Plan to Share IPD: Undecided